CLINICAL TRIAL: NCT00063141
Title: Revised Protocol 07 to Protocol CA225006 - A Phase III Randomized, Open-Label, Multicenter Study of Irinotecan and Cetuximab vs. Irinotecan as Second-Line Treatment in Patients With Metastatic, EGFR-Positive Colorectal Carcinoma
Brief Title: Study of Irinotecan and Cetuximab Versus Irinotecan as Second-Line Treatment in Patients With Metastatic, EGFR-Positive Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Chief Medical Officer, ImClone Systems
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA225-006; NCT00065598 (obsolete NCT alias)
Record Dates: First submitted 2003-06-20; First posted 2003-06-25 (Estimated); Last update posted 2010-04-12 (Estimated); Status verified 2010-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Irinotecan

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: cetuximab; Drug: Irinotecan
- Arm B (Active Comparator)
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: cetuximab — Vial, IV, 400 mg/m² week 1 then 250 mg/m², weekly, until PD/Toxicity/Pt-PI Decision
  Other Names: Erbitux
  Arms: Arm A
Drug: Irinotecan — Vial, IV, 350 mg/m², Q 3 Weeks, Until PD/Toxicity/Pt-PI Decision
  Arms: Arm A
Drug: Irinotecan — Vial, IV, 350 mg/m², Q 3 Weeks, Until PD/Toxicity/Pt-PI Decision
  Arms: Arm B

SUMMARY:
The purpose of this study is to determine whether overall survival is prolonged in subjects with metastatic, epidermal growth factor receptor (EGFR)-positive colorectal cancer treated with cetuximab in combination with irinotecan compared with irinotecan alone as second-line therapy following treatment with a fluoropyrimidine and oxaliplatin based, non-irinotecan-containing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented colorectal cancer which is EGFR-positive by immunohistochemistry [IHC] (may be based on archival samples) and is metastatic.
* Prior oxaliplatin administered for the first-line treatment of metastatic colorectal cancer.
* Prior fluoropyrimidine-containing regimen (5-fluorouracil [5-FU], capecitabine, or uracil/tegafur [UFT]), for the first-line treatment of metastatic disease.

Exclusion Criteria:

* A serious uncontrolled medical disorder that, in the opinion of the Investigator, would impair the ability of the subject to receive protocol therapy
* Unresolved diarrhea, bowel obstruction, or history of inflammatory bowel disease
* Known or documented brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1302 (Actual)
Dates: Start 2003-04; Primary Completion 2006-06 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Every 3 months after subject off-treatment

SECONDARY OUTCOMES:
Progression Free Survival | Q6 Weeks
Response | Q6 Weeks
Duration of Response | Q6 Weeks
Time to Response | Q6 Weeks
Disease Control Rate | Q6 Weeks
Safety | Q3 Weeks
Quality of Life | Q6 Weeks
Health Economics | Q3 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: E-mail: ClinicalTrials@ ImClone.com, Study Chair — Eli Lilly and Company
Locations (179):
- United States (107):
  - ImClone Investigational Site, Tucson, Arizona
  - ImClone Investigational Site, Pine Bluff, Arkansas
  - ImClone Investigational Site, Bakersfield, California
  - ImClone Investigational Site, Berkeley, California
  - ImClone Investigational Site, Beverly Hills, California
  - ImClone Investigational Site, Corona, California
  - ImClone Investigational Site, Gilroy, California
  - ImClone Investigational Site, Greenbrae, California
  - ImClone Investigational Site, Long Beach, California
  - ImClone Investigational Site, Los Angeles, California
  - ImClone Investigational Site, Montebello, California
  - ImClone Investigational Site, Orange, California
  - ImClone Investigational Site, Palm Springs, California
  - ImClone Investigational Site, Rancho Mirage, California
  - ImClone Investigational Site, San Diego, California
  - ImClone Investigational Site, Stockton, California
  - ImClone Investigational Site, Vallejo, California
  - ImClone Investigational Site, Aurora, Colorado
  - ImClone Investigational Site, Denver, Colorado
  - ImClone Investigational Site, New Haven, Connecticut
  - ImClone Investigational Site, New London, Connecticut
  - ImClone Investigational Site, Norwich, Connecticut
  - ImClone Investigational Site, Stamford, Connecticut
  - ImClone Investigational Site, Fort Myers, Florida
  - ImClone Investigational Site, Inverness, Florida
  - ImClone Investigational Site, Jacksonville, Florida
  - ImClone Investigational Site, Lakeland, Florida
  - ImClone Investigational Site, Miami, Florida
  - ImClone Investigational Site, New Port Richey, Florida
  - ImClone Investigational Site, Orlando, Florida
  - ImClone Investigational Site, Port Saint Lucie, Florida
  - ImClone Investigational Site, Atlanta, Georgia
  - ImClone Investigational Site, Columbus, Georgia
  - ImClone Investigational Site, Macon, Georgia
  - ImClone Investigational Site, Savannah, Georgia
  - ImClone Investigational Site, Tucker, Georgia
  - ImClone Investigational Site, Honolulu, Hawaii
  - ImClone Investigational Site, Naperville, Illinois
  - ImClone Investigational Site, South Bend, Indiana
  - ImClone Investigational Site, Kansas City, Kansas
  - ImClone Investigational Site, Overland Park, Kansas
  - ImClone Investigational Site, Lexington, Kentucky
  - ImClone Investigational Site, Louisville, Kentucky
  - ImClone Investigational Site, Richmond, Kentucky
  - ImClone Investigational Site, Baton Rouge, Louisiana
  - ImClone Investigational Site, Lafayette, Louisiana
  - ImClone Investigational Site, Metairie, Louisiana
  - ImClone Investigational Site, Shreveport, Louisiana
  - ImClone Investigational Site, Baltimore, Maryland
  - ImClone Investigational Site, Frederick, Maryland
  - ImClone Investigational Site, Boston, Massachusetts
  - ImClone Investigational Site, Ann Arbor, Michigan
  - ImClone Investigational Site, Detroit, Michigan
  - ImClone Investigational Site, Southfield, Michigan
  - ImClone Investigational Site, Minneapolis, Minnesota
  - ImClone Investigational Site, Robbinsdale, Minnesota
  - ImClone Investigational Site, Saint Louis Park, Minnesota
  - ImClone Investigational Site, Jackson, Mississippi
  - ImClone Investigational Site, Kansas City, Missouri
  - ImClone Investigational Site, Rolla, Missouri
  - ImClone Investigational Site, St Louis, Missouri
  - ImClone Investigational Site, Trenton, New Jersey
  - ImClone Investigational Site, Voorhees Township, New Jersey
  - ImClone Investigational Site, Albany, New York
  - ImClone Investigational Site, East Setauket, New York
  - ImClone Investigational Site, Latham, New York
  - ImClone Investigational Site, Mineola, New York
  - ImClone Investigational Site, New York, New York
  - ImClone Investigational Site, Rexford, New York
  - ImClone Investigational Site, Stony Brook, New York
  - ImClone Investigational Site, The Bronx, New York
  - ImClone Investigational Site, Valhalla, New York
  - ImClone Investigational Site, Durham, North Carolina
  - ImClone Investigational Site, Greenville, North Carolina
  - ImClone Investigational Site, High Point, North Carolina
  - ImClone Investigational Site, Raleigh, North Carolina
  - ImClone Investigational Site, Winston-Salem, North Carolina
  - ImClone Investigational Site, Bismarck, North Dakota
  - ImClone Investigational Site, Cincinnati, Ohio
  - ImClone Investigational Site, Cleveland, Ohio
  - ImClone Investigational Site, Columbus, Ohio
  - ImClone Investigational Site, Dayton, Ohio
  - ImClone Investigational Site, Newark, Ohio
  - ImClone Investigational Site, Oklahoma City, Oklahoma
  - ImClone Investigational Site, Hershey, Pennsylvania
  - ImClone Investigational Site, Philadelphia, Pennsylvania
  - ImClone Investigational Site, Pittsburgh, Pennsylvania
  - ImClone Investigational Site, Greenville, South Carolina
  - ImClone Investigational Site, Knoxville, Tennessee
  - ImClone Investigational Site, Memphis, Tennessee
  - ImClone Investigational Site, Nashville, Tennessee
  - ImClone Investigational Site, Austin, Texas
  - ImClone Investigational Site, Dallas, Texas
  - ImClone Investigational Site, Houston, Texas
  - ImClone Investigational Site, Plano, Texas
  - ImClone Investigational Site, Temple, Texas
  - ImClone Investigational Site, Ogden, Utah
  - ImClone Investigational Site, Arlington, Virginia
  - ImClone Investigational Site, Danville, Virginia
  - ImClone Investigational Site, Newport News, Virginia
  - ImClone Investigational Site, Richmond, Virginia
  - ImClone Investigational Site, Seattle, Washington
  - ImClone Investigational Site, Spokane, Washington
  - ImClone Investigational Site, Walla Walla, Washington
  - ImClone Investigational Site, Green Bay, Wisconsin
  - ImClone Investigational Site, Madison, Wisconsin
  - ImClone Investigational Site, Milwaukee, Wisconsin
- Australia (7):
  - ImClone Investigational Site, Perth, Australian Capital Territory
  - ImClone Investigational Site, Sydney, Australian Capital Territory
  - ImClone Investigational Site, Sydney, New South Wales
  - ImClone Investigational Site, Wollongong, New South Wales
  - ImClone Investigational Site, South Brisbane, Queensland
  - ImClone Investigational Site, Adelaide, South Australia
  - ImClone Investigational Site, Wien
- Austria (4):
  - ImClone Investigational Site, Graz
  - ImClone Investigational Site, Salzburg
  - ImClone Investigational Site, Vienna
  - ImClone Investigational Site, Wein
- ImClone Investigational Site, Charleroi, Belgium
- Czechia (3):
  - ImClone Investigational Site, Brno
  - ImClone Investigational Site, Olomouc
  - ImClone Investigational Site, Prague
- ImClone Investigational Site, Helsinki, Finland
- France (4):
  - ImClone Investigational Site, Avignon
  - ImClone Investigational Site, Marseille
  - ImClone Investigational Site, Nice
  - ImClone Investigational Site, Saint-Herblain
- Germany (18):
  - ImClone Investigational Site, Aschaffenburg
  - ImClone Investigational Site, Augsburg
  - ImClone Investigational Site, Dessau
  - ImClone Investigational Site, Dortmund
  - ImClone Investigational Site, Essen
  - ImClone Investigational Site, Hamburg
  - ImClone Investigational Site, Hanburg
  - ImClone Investigational Site, Kaiserslautern
  - ImClone Investigational Site, Kassel
  - ImClone Investigational Site, Magdeburg
  - ImClone Investigational Site, Mainz
  - ImClone Investigational Site, Mannheim
  - ImClone Investigational Site, Muchnhen
  - ImClone Investigational Site, München
  - ImClone Investigational Site, Regensburg
  - ImClone Investigational Site, Saarbrücken
  - ImClone Investigational Site, Stralsund
  - ImClone Investigational Site, Stuttgart
- ImClone Investigational Site, Hong Kong, Hong Kong
- Italy (14):
  - ImClone Investigational Site, Rozzano, Milano
  - ImClone Investigational Site, Ancona
  - ImClone Investigational Site, Bergamo
  - ImClone Investigational Site, Candiolo
  - ImClone Investigational Site, Florence
  - ImClone Investigational Site, Genova
  - ImClone Investigational Site, Livomo
  - ImClone Investigational Site, Milan
  - ImClone Investigational Site, Modena
  - ImClone Investigational Site, Napoli
  - ImClone Investigational Site, Perugia
  - ImClone Investigational Site, Reggio Emilia
  - ImClone Investigational Site, Roma
  - ImClone Investigational Site, Rome
- Netherlands (2):
  - ImClone Investigational Site, Apeldoorn
  - ImClone Investigational Site, Dordrecht
- Norway (2):
  - ImClone Investigational Site, Montebello, Oslo County
  - ImClone Investigational Site, Oslo
- ImClone Investigational Site, Porto, Portugal
- ImClone Investigational Site, Bratislava, Slovakia
- Sweden (2):
  - ImClone Investigational Site, Lund
  - ImClone Investigational Site, Stockholm
- Switzerland (3):
  - ImClone Investigational Site, Bern
  - ImClone Investigational Site, Liestal
  - ImClone Investigational Site, Zurich
- United Kingdom (8):
  - ImClone Investigational Site, Foresterhill, Aberdeenshire
  - ImClone Investigational Site, Hull, Avon
  - ImClone Investigational Site, Glasgow, Central
  - ImClone Investigational Site, Poole, Dorset
  - ImClone Investigational Site, London, Greater London
  - ImClone Investigational Site, Bournemouth, Hampshire
  - ImClone Investigational Site, Guildford, Surrey
  - ImClone Investigational Site, Sutton, Surrey